CLINICAL TRIAL: NCT06100146
Title: Does Small Scale Cereal-based Fortification Hold the Key to Improved Micronutrient Status in Ethiopia? The Case of Folic Acid and Vitamin B12 in Teenage Girls in Arba Minch, Ethiopia
Brief Title: Effectiveness of Fortification With Folic Acid and Vitamin B12 Among Teenage Girls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Collaborators: Arba Minch University (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Addis Ababa University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ONZ-2023-0137-C
Record Dates: First submitted 2023-10-03; First posted 2023-10-25 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Folate Deficiency; Vitamin B 12 Deficiency; Anemia, Megaloblastic; Cognitive Development; Depressive Symptoms
Keywords: Small scale fortification; Folic acid; Vitamin B12; Anemia; Cognitive development; Teenage girls
MeSH Terms: conditions — Folic Acid Deficiency; Vitamin B 12 Deficiency; Anemia, Megaloblastic; Depression; Anemia | interventions — Folic Acid; Control Groups

STUDY DESIGN:
Intervention Model Description: In randomized control trial, eligible teenage girls attending one of the schools in AM-HDSS will be randomly assigned to:
  1. An intervention group receiving a standard bag of cereal flours fortified with folic acid and Vitamin B12 at local mills every week for six months.
  2. A placebo group receiving a standard bag of unfortified cereal flours every week for six months.
  Participants in all the treatment groups remain eligible to benefit from the standard health care and nutrition programs provided at school, such as deworming at the beginning of the school year.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Flours will be indistinguishable in appearance except for the vitamins added to the flours of the intervention group. An independent trained person will be assigned to monitor the fortification process and the two products will be packed immediately and coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Teenage girls randomly assigned to the control group will receive a standard bag of unfortified cereal flours every week for six months.
  Interventions: Other: Unfortified cereal flour
- folic acid & vit B12 fortified flour (Experimental): Teenage girls randomly assigned to the control group will receive a standard bag of cereal flours fortified with folic acid and Vit B12 every week for six months.
  Interventions: Dietary Supplement: Folic acid and vitamin B12 fortified flour

INTERVENTIONS:
Dietary Supplement: Folic acid and vitamin B12 fortified flour — Standard bags of fortified cereal-based flours will be prepared at local mills from the common staple cereal food in the area. The dose of vitamins will be added to the flour of the intervention group and mixed with batch mixing technique. The concentration of folic acid and vitamin B12 per 1kg of flour will be 2mg and 0.02mg, respectively. Participants will be supplied with 6 kg bags of flour, which will be enough for 30 days, and 1.5kg bags of flour will be delivered to their home on a weekly basis and lasting for 6 months. Instructions on the preparation of meals and frequency of intake with a weekly compliance sheet will be provided for monitoring the intervention.
  Other Names: Intervention group
  Arms: folic acid & vit B12 fortified flour
Other: Unfortified cereal flour — Standard bags of unfortified cereal-based flours will be prepared at local mills from the common staple cereal food in the area. Participants will be supplied with 6 kg bags of flour, which will be enough for 30 days, and 1.5kg bags of flour will be delivered to their home on a weekly basis and lasting for 6 months. Instructions on the preparation of meals and frequency of intake with a weekly compliance sheet will be provided for monitoring the intervention.
  Other Names: Control group
  Arms: Control group

SUMMARY:
Folic acid and vitamin B12 play an interdependent role in key cellular processes, namely deoxyribonucleic acid synthesis, cell division, red blood cell formation, and nervous system myelination. A deficiency of either vitamin will predispose teenagers to many diseases, which persist across their lifespan. Fortification of food with micronutrients has been promoted to reduce micronutrient deficiencies. A large segment of vulnerable populations in low- and middle-income countries (LMICs) resides in rural settings and has limited access to large-scale commercialized fortified foods. In such operational constraints, the use of locally (small-scale) fortified cereals could be an alternative intervention. The study aims to evaluate the effectiveness of small scale folic acid and vitamin B12 fortified cereals in improving folate and vitamin B12 status, growth velocity, puberty status, anaemia, cognitive development and mental health among teenage girls, in rural rift valley of Ethiopia.

DETAILED DESCRIPTION:
Folic acid (FA) and vitamin B12 play an interdependent role in key cellular processes, namely deoxyribonucleic acid synthesis, cell division, red blood cell formation, and nervous system myelination. Teenagers are the future mothers. Hence their health and nutritional status have long term consequences on future pregnancies and birth outcomes. Neural Tube Defects (NTDs) are a group of fatal or severely disabling birth defects known to be mainly a consequence of severe folate deficiency in early pregnancy. The policy of advising women to take iron & FA (IFA) supplements during pregnancy has not been successful in preventing NTDs because of the low adherence to antenatal care services including IFA, the large proportion of unplanned pregnancies, the timing at which IFA supplementation starts, and the logistical limitation that makes the access to IFA limited. The evidence is strong on the importance of food fortification in the promotion of maternal and child health mainly through reducing micronutrient deficiencies. A large segment of vulnerable populations in developing countries resides in rural settings and has limited access to fortified foods in the market. In such operational constraints, using locally fortified cereals could be an alternative intervention. However, there is a paucity of evidence regarding effectiveness of small-scale cereal-based fortification; in Ethiopia, the evidence is inexistent. Moreover, teenage girls are an under-studied group and do not constitute a target population from different nutritional intervention programs.

The overall objective of this study is to evaluate the effectiveness of small-scale folic acid and vitamin B12-fortified cereals in improving folate and vitamin B12 status, growth velocity, puberty status, anaemia, cognitive development and mental health among rural teenage girls (13-19 years of age).

This study will be conducted in Arba Minch Health and Demographic Surveillance Sites (AM-HDSS), Southern Ethiopia from October 2023 to April 2024. Effectiveness of intake of folic acid and vitamin B12 fortified meals will be evaluated in a randomized, double-blind controlled trial among 474 teenage girls between 13 and 19 years of age who are residing in and attending one of the schools at AM-HDSS.

Data on the following variables, except for demographic characteristics of teenage girls and their respective parents and/or household heads will be collected at the start and end point of the 6 months intervention. Data collection will be carried out at schools and at respective girls' home.

* Demographic characteristics of the teenage girls, morbidity status, helminthic infections, dietary intake, anthropometry, puberty status, presence of depressive symptoms, biochemical samples and cognitive development will be assessed in teenage girls directly at schools.
* Socio-demographic characteristics of the parents or the head of the household if different from parents, family wealth status, food security, health care services and environmental characteristics will be collected in recruited teenage girls' households within the one week following the enrolment and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Teenage girls between 13 and 19 years of age who live in households at Arba Minch Health and Demographic Surveillance Sites (AM-HDSS) are eligible to participate in the study if:

* One or both of their parents signed an informed consent form and the girl's agreement.
* Their parents and the girl planned to stay in the study area during the period of the study (minimum 6 months) in the kebele.
* Both parents and girls accept the intervention packages including blood draws and home visits.

Exclusion Criteria:

* Chronically ill girls diagnosed with diabetes and asthma;
* Severely undernourished girls (defined as body mass index z score < -3 standard deviations of the median World Health Organization reference population);
* Severely anaemic girls (Hb concentration <80g/L);
* Teenage girls who are pregnant, lactating or taking IFA/B12 supplements;
* Diagnosed hemoglobinopathy (sickle cell or thalassemia);
* Diagnosed liver diseases like acute hepatitis, cirrhosis, hepatocellular carcinoma, and metastatic liver disease

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 474 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum folic acid concentrations | Assessed at 6 months
  Serum folate levels ng/ml (nmol/l)
Erythrocyte (RBC) folic acid concentrations | Assessed at 6 months
  RBC folate level ng/ml (nmol/l)
General cognitive ability | Assessed at 6 months
  Raven Progressive Matrices (RPM) tests, a measure of nonverbal intelligence.
Working memory | Assessed at 6 months
  Digit Span (Forward, Backward, and Sequencing) is a standardized test that assesses the working memory of participants.
Depression | Assessed at 6 months
  Depressive symptoms will be assessed by Patient Health Questionnaire (PHQ) 9 modified for adolescents (PHQ-9A), a self-report instrument comprised of 9-items. Items are rated on a four-point ordinal scale.
Serum vitamin B12 concentrations | Assessed at 6 months
  Serum vitamin B12 level (pmol/L)
Fat-free mass | Assessed at 6 months
  An index of adiposity will be measured to evaluate girls' body composition, in %
Fat mass | Assessed at 6 months
  An index of adiposity will be measured to evaluate girls' body composition, in kg

SECONDARY OUTCOMES:
RBC structure (megaloblastic anaemia) | Assessed at 6 months
  Mean Corpuscular Volume (MCV) in femtoliters/fl
Plasma homocysteine concentrations | Assessed at 6 months
  Plasma homocysteine level (µmol/L)
Weight | Assessed at 3 and 6 months
  Participant weight (kg)
Adherence to the intervention/fortification | Assessed weekly for the whole period of intervention (until 6 months)
  adherence to the flour consumption will be assessed through home to home visit in a weekly basis.
Haemoglobin concentration | Assessed at 6 months
  Haemoglobin concentration (g/dl)
Height | Assessed at 6 months
  Participant height (cm)
Puberty status | Assessed at 6 months of fortification
  The pubertal status will be assessed by Pubertal Development Scale which has a 4-point scale ranging from 1 (has not begun) to 4 (development completed). Girls will report on their body hair development, growth spurt, skin changes, breast development and the occurrence of menarche (1=no and 4=yes).
Prevalence of soil-transmitted helminths | Assessed at 6 months
  The presence of worm parasites and egg density in the stools. Three common parasites and their eggs will be investigated, i.e. Ascaris lumbricoides (round worm), Trichuris trichiura (whipworm) and Ancyclostoma duodenale or Necater americanus (hookworms)
Prevalence of Schistosome infection | Assessed at 6 months
  The prevalence of Schistosoma mansoni infection

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, MD,PHD, Principal Investigator — University Ghent
Locations (2):
- Ethiopia (2):
  - Arba Minch Health and Demographic Surveillance System sites, Arba Minch
  - Arba Minch University, Arba Minch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oumer M, Taye M, Aragie H, Tazebew A. Prevalence of Spina Bifida among Newborns in Africa: A Systematic Review and Meta-Analysis. Scientifica (Cairo). 2020 Oct 6;2020:4273510. doi: 10.1155/2020/4273510. eCollection 2020. PMID 33083093
- [Background] Wald NJ. Postscript to 'Folic acid and neural tube defects: Discovery, debate and the need for policy change'. J Med Screen. 2022 Sep;29(3):147. doi: 10.1177/09691413221117464. Epub 2022 Aug 8. No abstract available. PMID 35942520
- [Background] Ardila A. Development of metacognitive and emotional executive functions in children. Appl Neuropsychol Child. 2013;2(2):82-7. doi: 10.1080/21622965.2013.748388. Epub 2013 Jan 28. PMID 23848243
- [Background] Centeno Tablante E, Pachon H, Guetterman HM, Finkelstein JL. Fortification of wheat and maize flour with folic acid for population health outcomes. Cochrane Database Syst Rev. 2019 Jul 1;7(7):CD012150. doi: 10.1002/14651858.CD012150.pub2. PMID 31257574
- [Background] Mildon A, Klaas N, O'Leary M, Yiannakis M. Can fortification be implemented in rural African communities where micronutrient deficiencies are greatest? Lessons from projects in Malawi, Tanzania, and Senegal. Food Nutr Bull. 2015 Mar;36(1):3-13. doi: 10.1177/156482651503600101. PMID 25898711